CLINICAL TRIAL: NCT04121273
Title: Clinical Study of GPC3-targeted Chimeric Antigen Receptor T Cells fo Treating Advanced Hepatocellular Carcinoma
Brief Title: GPC3-targeted CAR-T Cell for Treating GPC3 Positive Advanced HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Beicheng Sun, Director of Hepatobiliary Surgery, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v1.0 20180620
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: chimeric antigen receptor T cell (CAR- T); glypican-3 (GPC3); hepatocellular carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Simpson-Golabi-Behmel syndrome | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells (Experimental): CAR-T cells targeting GPC3 will be administered to enrolled patients with hepatocellular carcinoma.
  Interventions: Biological: CAR-T cell immunotherapy

INTERVENTIONS:
Biological: CAR-T cell immunotherapy — Patients enrolled will recieve three different doses of the CAR-T cell every two weeks as follows:
  Dose 1: 1x10^7/m2
  Dose 2: 3x10^7/m2
  Dose 3: 1x10^8/m2
  The cell numbers are calculated according to CAR-positive T cells.

SUMMARY:
Patients with hepatocellular carcinoma (a type of primary liver cancers) are enrolls in this study. The cancer has progressed after standard treatment, or the patient cannot receive regular treatment.

Investigator made a gene called chimeric antigen receptor derived from an antibody that recognizes Glypican 3, a protein detected in in a large proportion of hepatocellular carcinoma. The gene will introduce into T cell from patient's blood to make them recognize and kill cancer cells.

The aim of this study is to evaluate the efficacy, tolerance and safety of chimeric antigen receptor-modified T (CAR-T) cell targeting Glypican 3 for advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. GPC3 positive HCC, tumor size >= 5 cm, cannot receive standard treatment, Expected survival time>=3 months.
2. Routine blood test: white blood cell count（WBC)>= 2.5×10^9/L, hemoglobin (Hb)>= 9.0 g/dL, blood platelet >= 60×10^9/L, Lymphocyte percentage>=15%.
3. Blood biochemical parameters: ALB >= 30 g/L, ALT <= 5 times of the normal value, AST <= 5 times of the normal value, serum lipase<=1.5 times of the normal value, serum amylase<=1.5 times of the normal value， total bilirubin <= 2.5 times of the normal value.
4. Prothrombin time INR < 1.7.
5. Ejection fraction (EF) >= 55%, oxygen saturation (SO2) > 90%.
6. No allergic reaction to contrast material.
7. Karnofsky score >= 60%.
8. Child-puge score <7.
9. Peripheral venous access.
10. Voluntarily signed informed consent.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Systemic steroid treatment ( >prednisone equivalent/kg/day).
3. Patients with previous history of cell immunotherapy or antibody therapy.
4. Patients received radiotherapy/chemotherapy in the past 4 weeks.
5. Patients are participating in other clinical trials.
6. Patients with uncontrolled symptoms including infection, heart failure, arrhythmia.
7. Patients with acute allergic reaction.
8. History of liver transplantation.
9. Patients with anticoagulant treatment.
10. Patients with hepatic encephalopathy.
11. Eligible for hepatectomy, liver transplantation or other standard treatment.
12. Unstable gastrointestinal and respiratory bleeding.
13. Active viral, fungal or bacterial infections.
14. Heart failure classification (NYHA): II-IV.
15. Patients are unable or unwilling to comply with the requirements of the study protocol.
16. Patients do not meet the criteria above.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-05 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patient with dose limiting toxicity | 2 months
  After each dose of T cell infusion, the adverse effects related to T cell therapy such as fever and jaundice are observed.

SECONDARY OUTCOMES:
Radiological evaluation of tumor size after CAR- T immunotherapy | 3 months
  Evaluate the therapeutic effect of CAR-T immunotherapy radiological observation of the tumor size after infusion of CAR-T cells.
Peripheral tumor marker | 3 months
  After CAR-T cell infusion, alpha fetoprotein (AFP) will be tested regularly in blood.
Number of Peripheral CAR-T cell | 3 months
  The number and proliferation in vivo are tested with Flow Cytometry regularly.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No